CLINICAL TRIAL: NCT05457959
Title: A Placebo-Controlled, Single (Participant) Blind Trial to Evaluate the Safety, Tolerability, and Early Immunogenicity of Peptide-Pulsed Dendritic Cell Vaccination With Nivolumab and Ipilimumab in Recurrent and/or Progressive Diffuse Hemispheric Glioma, H3 G34-Mutant
Brief Title: Peptide-Pulsed Dendritic Cell Vaccination in Combination With Nivolumab and Ipilimumab for the Treatment of Recurrent and/or Progressive Diffuse Hemispheric Glioma, H3 G34-mutant
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Never opened
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 22-000581; NCI-2022-05326 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-07-07; First posted 2022-07-14 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-03

CONDITIONS: Diffuse Hemispheric Glioma, H3 G34-Mutant
MeSH Terms: interventions — Ipilimumab; CTLA-4 Antigen; Leukapheresis; Nivolumab; poly ICLC

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort I Arm A (ppDC, placebo) (Placebo Comparator): Patients undergo leukapheresis 10 days prior to first injection. Patients receive ppDC ID in both arms with poly ICLC IM on day -10 and placebo IV on day -9 prior to standard of care surgical resection.
  Interventions: Biological: Dendritic Cell Tumor Peptide Vaccine; Procedure: Leukapheresis; Drug: Placebo Administration; Drug: Poly ICLC; Procedure: Resection
- Cohort I Arm B (placebo, nivolumab, ipilimumab) (Placebo Comparator): Patients undergo leukapheresis 10 days prior to first injection. Patients receive placebo ID in both arms with poly ICLC IM on day -10 and nivolumab IV and ipilimumab IV on day -9 prior to standard of care surgical resection.
  Interventions: Biological: Ipilimumab; Procedure: Leukapheresis; Biological: Nivolumab; Drug: Placebo Administration; Drug: Poly ICLC; Procedure: Resection
- Cohort I Arm C (ppDC, nivolumab, ipilimumab) (Experimental): Patients undergo leukapheresis 10 days prior to first injection. Patients receive ppDC ID divided in both arms with poly ICLC IM on day -10 and nivolumab IV and ipilimumab IV on day -9 prior to standard of care surgical resection.
  Interventions: Biological: Dendritic Cell Tumor Peptide Vaccine; Biological: Ipilimumab; Procedure: Leukapheresis; Biological: Nivolumab; Drug: Poly ICLC; Procedure: Resection
- Cohort II Arm A (ppDC, placebo) (Experimental): Within 30 days of surgical resection, patients receive ppDC ID in both arms with poly ICLC IM and placebo IV on day 1 of each cycle. Treatment repeats every 2 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Post-treatment, patients may receive nivolumab IV on day 1 of each cycle. Cycles repeat every 4 weeks for up to 24 months following surgical resection in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Dendritic Cell Tumor Peptide Vaccine; Drug: Placebo Administration; Drug: Poly ICLC
- Cohort II Arm B (placebo, nivolumab) (Placebo Comparator): Within 30 days of surgical resection, patients receive placebo ID in both arms with poly ICLC IM and nivolumab IV on day 1 of each cycle. Treatment repeats every 2 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Post-treatment, patients may receive nivolumab IV on day 1 of each cycle. Cycles repeat every 4 weeks for up to 24 months following surgical resection in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Drug: Placebo Administration; Drug: Poly ICLC
- Cohort II Arm C (ppDC, nivolumab) (Experimental): Within 30 days of surgical resection, patients receive ppDC ID in both arms with poly ICLC IM and nivolumab IV on day 1 of each cycle. Treatment repeats every 2 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Post-treatment, patients may receive nivolumab IV on day 1 of each cycle. Cycles repeat every 4 weeks for up to 24 months following surgical resection in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Dendritic Cell Tumor Peptide Vaccine; Biological: Nivolumab; Drug: Poly ICLC

INTERVENTIONS:
Biological: Dendritic Cell Tumor Peptide Vaccine — Given ID
  Other Names: DC tumor peptide vaccine; dendritic cells pulsed with tumor peptide
  Arms: Cohort I Arm A (ppDC, placebo); Cohort I Arm C (ppDC, nivolumab, ipilimumab); Cohort II Arm A (ppDC, placebo); Cohort II Arm C (ppDC, nivolumab)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
  Arms: Cohort I Arm B (placebo, nivolumab, ipilimumab); Cohort I Arm C (ppDC, nivolumab, ipilimumab)
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
  Arms: Cohort I Arm A (ppDC, placebo); Cohort I Arm B (placebo, nivolumab, ipilimumab); Cohort I Arm C (ppDC, nivolumab, ipilimumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
  Arms: Cohort I Arm B (placebo, nivolumab, ipilimumab); Cohort I Arm C (ppDC, nivolumab, ipilimumab); Cohort II Arm B (placebo, nivolumab); Cohort II Arm C (ppDC, nivolumab)
Drug: Placebo Administration — Given ID
  Arms: Cohort I Arm B (placebo, nivolumab, ipilimumab); Cohort II Arm B (placebo, nivolumab)
Drug: Placebo Administration — Given IV
  Arms: Cohort I Arm A (ppDC, placebo); Cohort II Arm A (ppDC, placebo)
Drug: Poly ICLC — Given IM
  Other Names: Hiltonol; Poly I:Poly C with Poly-L-Lysine Stabilizer; poly-ICLC; PolyI:PolyC with Poly-L-Lysine Stabilizer; Polyinosinic-Polycytidylic Acid Stabilized with Polylysine and Carboxymethylcellulose; Polyriboinosinic-Polyribocytidylic Acid-Polylysine Carboxymethylcellulose; Stabilized Polyriboinosinic/Polyribocytidylic Acid
Procedure: Resection — Undergo standard of care surgical resection
  Other Names: Surgical Resection
  Arms: Cohort I Arm A (ppDC, placebo); Cohort I Arm B (placebo, nivolumab, ipilimumab); Cohort I Arm C (ppDC, nivolumab, ipilimumab)

SUMMARY:
This phase I trial tests peptide-pulsed dendritic cell vaccination in combination with immunotherapy nivolumab and ipilimumab for the treatment diffuse hemispheric glioma with a H3 G34 mutation that has come back (recurrent) and/or is growing, spreading, or getting worse (progressive). Vaccines made from the patient's own white blood cells and peptide-pulsed dendritic cells may help the body build an effective immune response to kill tumor cells. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, also may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Together, the vaccine and immunotherapy drugs given before and after surgical resection (the removal of tumor cells through surgery) may improve stimulation of anti-tumor immunity to help fight the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of nivolumab/ipilimumab and peptide-pulsed dendritic cell (ppDC) vaccination in diffuse hemispheric glioma H3 G34-mutant (DHG) participants undergoing surgical resection.

SECONDARY OBJECTIVES:

I. To determine whether nivolumab/ipilimumab and/or ppDC vaccination facilitate intratumoral T cell-mediated anti-tumor immune activation in progressive DHG.

II. To determine whether nivolumab/ipilimumab and/or ppDC vaccination stimulate systemic adaptive anti-tumor immunity in progressive DHG.

OUTLINE: Patients are sequentially assigned to 2 cohorts.

COHORT 1 (Pre-Surgical Resection): Patients are randomized to 1 of 3 arms.

ARM A: Patients undergo leukapheresis 10 days prior to first injection. Patients receive ppDC intradermally (ID) in both arms with poly ICLC intramuscularly (IM) on day -10 and placebo intravenously (IV) on day -9 prior to standard of care surgical resection.

ARM B: Patients undergo leukapheresis 10 days prior to first injection. Patients receive placebo ID in both arms with poly ICLC IM on day -10 and nivolumab IV and ipilimumab IV on day -9 prior to standard of care surgical resection.

ARM C: Patients undergo leukapheresis 10 days prior to first injection. Patients receive ppDC ID divided in both arms with poly ICLC IM on day -10 and nivolumab IV and ipilimumab IV on day -9 prior to standard of care surgical resection.

COHORT 2 (Post-Surgical Resection): Patients are assigned to 1 of 3 arms.

ARM A: Within 30 days of surgical resection, patients receive ppDC ID in both arms with poly ICLC IM and placebo IV on day 1 of each cycle. Treatment repeats every 2 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Post-treatment, patients may receive nivolumab IV on day 1 of each cycle. Cycles repeat every 4 weeks for up to 24 months following surgical resection in the absence of disease progression or unacceptable toxicity.

ARM B: Within 30 days of surgical resection, patients receive placebo ID in both arms with poly ICLC IM and nivolumab IV on day 1 of each cycle. Treatment repeats every 2 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Post-treatment, patients may receive nivolumab IV on day 1 of each cycle. Cycles repeat every 4 weeks for up to 24 months following surgical resection in the absence of disease progression or unacceptable toxicity.

ARM C: Within 30 days of surgical resection, patients receive ppDC ID in both arms with poly ICLC IM and nivolumab IV on day 1 of each cycle. Treatment repeats every 2 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Post-treatment, patients may receive nivolumab IV on day 1 of each cycle. Cycles repeat every 4 weeks for up to 24 months following surgical resection in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and 6 months and every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 13 and 60 years with pathologically-confirmed diagnosis of (or pathology re-review consistent with) DHG will be enrolled in this study
* All participants must be undergoing clinically indicated resection surgical resection with the goal of cytoreduction
* Participants must undergo human leukocyte antigen (HLA) testing
* A female participant who has childbearing potential must have negative urine or serum pregnancy test 72 hours prior to the first dose and be willing to use adequate method of contraception for course of study and 120 days after last dose
* The participant (or legally acceptable representative if applicable) provides informed consent (and written assent from minors) for the trial
* Have unequivocal evidence for contrast-enhancing tumor progression by modified response assessment in neuro-oncology (mRANO) criteria based on MRI scan within 72 days prior to enrollment. This criterion will be reviewed by investigators prior to enrollment
* An interval of the following durations prior to enrollment:

  * At least 14 days from prior surgical resection
  * At least 7 days from prior stereotactic biopsy
  * At least 12 weeks from prior radiotherapy, unless there is unequivocal histologic confirmation of tumor progression
  * At least 23 days from prior chemotherapy
  * At least 42 days from nitrosureas
* Have sufficient archival tumor tissue confirming high-grade glioma (HGG) or variants for submission following registration. The following amount of tissue is required: 1 formalin-fixed, paraffin embedded (FFPE) tissue block (preferred) or 10 FFPE unstained slides (5 um thick)
* Have a Karnofsky Performance Status (KPS) >= 70, if participant age >= 16. Have a Lansky Performance Status (LPS) >= 70, if participant age < 16
* Absolute neutrophil count (ANC) >= 1500/uL (within 14 days prior to start of study treatment)
* Platelets >= 100 000/uL (microliter) (within 14 days prior to the start of study treatment)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (within 14 days prior to the start of study treatment)

  * Note: Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (CrCl) >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) (within 14 days prior to the start of study treatment)

  * Note: Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (within 14 days prior to the start of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases) (within 14 days prior to the start of study treatment)
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants (within 14 days prior to the start of study treatment)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (within 14 days prior to the start of study treatment)

Exclusion Criteria:

* Age < 13 years or > 60 years
* Have had more than 2 separately-treated recurrences of the index tumor
* A woman of child-bearing potential who has a positive urine pregnancy test within 72 hours prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory target (e.g., CTLA-4, OX 40, CD137)
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to enrollment

  * Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline. Participants with =< grade 2 neuropathy may be eligible
  * Note: If participant received major surgical resection, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Has received prior radiotherapy within 12 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 12 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment

  * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Has a diagnosis of immunodeficiency or is receiving chronic systemic corticosteroid therapy (dosing exceeding 1 mg/kg/day of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years

  * Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has severe hypersensitivity (>= grade 3) to nivolumab or ipilimumab, and/or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (HCV) (defined as HCV ribonucleic acid (RNA) is detected) infection

  * Note: No testing for hepatitis B and hepatitis C is required unless mandated by local health authority
* Has a known history of active tuberculosis (bacillus tuberculosis)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Kidney dysfunction precluding administration of gadolinium-based contrast
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Start of treatment up to 100 days post-treatment
  Safety and tolerability will be monitored by the University of California, Los Angeles (UCLA) Data Safety Monitoring Board (DSMB) incorporating regular reviews with the investigators in this pilot surgical trial. Adverse events will be monitored throughout the trial and graded in severity according to the guidelines outlined in the Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

SECONDARY OUTCOMES:
Increased tumor-infiltrating lymphocyte (TIL) density | Up to 2 years
  Tumor tissue will be analyzed for increased TIL density, quantified as number of cytotoxic T lymphocytes (CTLs) per nucleated cell, or increased T cell activation/ decreased T cell exhaustion marker expression. Mean differences for all outcomes of interest will be estimated for (group A versus group B, group A versus C, and group B versus C). Sampling uncertainty in estimation will be reported using 95% Confidence Intervals. A two-sample t-test with Bonferroni adjustment will be performed to test each of these two hypotheses.
Oligoclonal T cell expansion | Up to 2 years
  Peripheral blood will be analyzed for oligoclonal T cell expansion by T cell receptor (TCR)VBeta sequencing. Mean differences for all outcomes of interest will be estimated for (group A versus group B, group A versus C, and group B versus C). Sampling uncertainty in estimation will be reported using 95% Confidence Intervals. A two-sample t-test with Bonferroni adjustment will be performed to test each of these two hypotheses.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony C Wang, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States